CLINICAL TRIAL: NCT00316680
Title: Study to Assess Immunogenicity and Safety of GlaxoSmithKline Biologicals' Kft's DTPw-HBV/Hib vs DTPwCSL-HBV/Hib Kft and vs Concomitant Administration of CSL's Triple Antigen and GlaxoSmithKline Biologicals' Hiberix, to Infants at 2, 4, 6 Months of Age, After a Birth Dose of Hepatitis B
Brief Title: Immuno & Safety Study With 2 Formulations of DTPw-HBV/HIB When Given at Birth With Hepatitis B at 2, 4 and 6 Mths.Age.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 104489
Record Dates: First submitted 2006-04-20; First posted 2006-04-21 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Haemophilus Influenzae Type b; Diphtheria; Tetanus; Hepatitis B; Whole Cell Pertussis
MeSH Terms: conditions — Haemophilus Infections; Diphtheria; Tetanus; Hepatitis B | interventions — Tetanus Toxoid; Hepatitis B Vaccines; HibTITER protein, Haemophilus influenzae

INTERVENTIONS:
Biological: Diphtheria, tetanus, pertussis, hepatitis B, Hib vaccine
  Other Names: Diphtheria; tetanus; pertussis; hepatitis B; Hib vaccine

SUMMARY:
A trial to characterize the immunogenicity of 2 different formulations of a vaccine from GSK Biologicals, including the following five antigens: diphtheria, tetanus, pertussis, hepatitis B and Haemophilus influenzae type b. A vaccine from Commonwealth Serum Laboratories (diphtheria, tetanus, pertussis) which is co-administered with Haemophilus influenzae type b vaccine will also be used as a comparator. Reactogenicity and safety of all vaccines will be assessed as well.

DETAILED DESCRIPTION:
"The study will be carried out in a partially double blind manner (i.e. double blind with respect to DTPwGöd-HBV/Hib Kft and DTPwCSL-HBV/Hib Kft groups and open with respect to CSL's Triple Antigen & Hib group). Subjects will be randomly allocated to one of the three following groups to receive:

* GSK Biologicals Kft's combined DTPwGöd-HBV/Hib Kft vaccine.
* GSK Biologicals Kft's combined DTPwCSL-HBV/Hib Kft vaccine.
* CSL's Triple Antigen + GSK Biologicals' Hib vaccines. There will be a specific follow-up of solicited local and general symptoms during 4 days after each vaccination and of unsolicited symptoms for 31 days after each vaccination. Serious adverse events reported during the study period will be recorded.

"

ELIGIBILITY:
Inclusion criteria

* Administration of one dose of hepatitis B vaccine at birth.
* A healthy male or female between, and including, 6 and 12 weeks of age at the time of the first DTPw vaccination.

Exclusion criteria

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days before the first vaccine dose or planned administration during the study period with the exception of oral polio vaccine hepatitis B vaccine for the Triple Antigen + Hib group.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required)
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Bacille Calmette-Guérin (BCG) vaccine given after the first 2 weeks of life.
* Previous vaccination against diphtheria, tetanus, pertussis and/or Hib/History of diphteria, tetanus, pertussis, hepatitis B and/ or hib disease.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288
Dates: Start 2006-03; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
GMC of anti-BPT Ab

SECONDARY OUTCOMES:
anti-HBs, anti-diphtheria, anti-tetanus, anti-BPT & anti-PRP conc. & GMCs; vaccine response to BPT
Solicited & unsolicited symptoms, SAEs "

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register